CLINICAL TRIAL: NCT00360854
Title: Phase I Studies of TARCEVA™ (ERLOTINIB HYDROCHLORIDE, OSI-774) as Single Agent in Children With Refractory and Relapsed Malignant Brain Tumors and in Combination With Irradiation in Newly Diagnosed Brain Stem Glioma
Brief Title: Erlotinib Alone or in Combination With Radiation Therapy in Treating Young Patients With Refractory or Relapsed Malignant Brain Tumors or Newly Diagnosed Brain Stem Glioma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000481539; CCLG-NAG-2005-09; ITCC-003; EU-20617; CCLG-CPP-05-07; ROCHE-MO18461; EUDRACT-2004-005247-10
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway and hypothalamic glioma; childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; childhood low-grade cerebral astrocytoma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood brain tumor; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood pineoblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Choroid Plexus Neoplasms | interventions — Erlotinib Hydrochloride; Amplified Fragment Length Polymorphism Analysis; Radiotherapy

INTERVENTIONS:
Drug: erlotinib hydrochloride
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: pharmacological study
Radiation: radiation therapy

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving erlotinib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of erlotinib when given alone or together with radiation therapy in treating young patients with refractory or relapsed malignant brain tumors or newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the maximum tolerated dose of single-agent erlotinib hydrochloride in pediatric patients with refractory or relapsed malignant brain tumors and in combination with radiotherapy in pediatric patients with newly diagnosed brain stem glioma.

Secondary

* Determine dose-limiting toxicities of these regimens.
* Define the safety profile of these regimens.
* Characterize the pharmacokinetic behavior of erlotinib hydrochloride in these patients.
* Evaluate the efficacy of these regimens.
* Correlate expression and mutations of epidermal growth factor receptor with treatment response.

OUTLINE: This is a multicenter, nonrandomized, open-label, dose-escalation study of erlotinib hydrochloride. Patients are assigned to 1 of 2 treatment groups according to disease.

* Group 1 (refractory or relapsed malignant brain tumors): Patients receive oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of erlotinib hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).

* Group 2 (newly diagnosed brain stem glioma): Patients receive oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 21 days in the absence of unacceptable toxicity or disease progression. Beginning on day 1, patients also undergo radiotherapy 5 days a week for 6 weeks .

Cohorts of 1-2 patients receive escalating doses of erlotinib hydrochloride until the MTD is determined. The MTD is defined as the dose resulting in 25% of patients experiencing DLT at 6 weeks.

Blood is collected for pharmacokinetic assessments and pharmacogenetic genotyping for analysis of enzyme polymorphisms. Tumor tissue may be assessed for epidermal growth factor receptor mutations.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Histologically or cytologically confirmed malignant brain tumor

    * Refractory to first-line therapy or relapsed after conventional therapy
    * No effective conventional therapy exists
  * Histologically confirmed brain stem glioma

    * Newly diagnosed disease
    * No pilocytic glioma
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2 OR Lansky play scale 50-100%

  * Patients with motor paresis due to disease are eligible
  * Neurological deficits must be stable for ≥ 1 week
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count > 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8 g/dL
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance ≥ 70 mL/min
* No other serious, uncontrolled illness
* No active infection
* No organ toxicity ≥ grade 2 except alopecia and neurological symptoms due to disease
* Must be able to take oral medication

  * Patients with newly diagnosed brain stem glioma with difficulty swallowing may be eligible
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of pulmonary dysfunction or pre-existing lung disease
* No myocardial infarction within the past year
* No severe cardiac pathology
* No significant ophthalmologic abnormality including, but not limited to, any of the following:

  * Severe dry eye syndrome
  * Keratoconjunctivitis sicca
  * Sjögren's syndrome
  * Severe exposure keratitis
  * Any other disorder likely to increase the risk of corneal epithelial lesions

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* More than 6 weeks since prior radiotherapy
* No concurrent warfarin
* No other concurrent anticancer or investigational agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-05

PRIMARY OUTCOMES:
Maximum tolerated dose of erlotinib hydrochloride when given alone and in combination with radiotherapy

SECONDARY OUTCOMES:
Dose-limiting toxicities
Safety
Pharmacokinetic behavior of erlotinib hydrocloride
Efficacy
Correlation of expression and mutations of epidermal growth factor receptor with treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Darren Hargrave, MD — Royal Marsden NHS Foundation Trust
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales